CLINICAL TRIAL: NCT04906980
Title: A Phase 2a, Randomized, Double-blind, Placebo-controlled Trial to Evaluate the Antiviral Activity, Safety and Tolerability, and Pharmacokinetics of JNJ-64281802 in Participants With Confirmed Dengue Fever
Brief Title: A Study of JNJ-64281802 in Participants With Confirmed Dengue Fever
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Feasibility of enrollment impacted by COVID
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108919; 64281802DNG2003 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2021-05-26; First posted 2021-05-28 (Actual); Results first posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-01

CONDITIONS: Dengue
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- JNJ-64281802 (Experimental): Participants will receive 2 initial loading doses of JNJ-64281802 up to Day 2, followed by a maintenance dose on Days 3, 4, and 5.
  Interventions: Drug: JNJ-64281802
- Placebo (Placebo Comparator): Participants will receive oral dose of matching placebo every 8 hour (q8h) and once daily on Day 4 and Day 5.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JNJ-64281802 — JNJ-64281802 will be administered orally.
  Arms: JNJ-64281802
Drug: Placebo — Matching placebo (PEG400) will be administered orally.
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the antiviral activity of JNJ-64281802 versus placebo in terms of reduction of dengue virus (DENV) ribonucleic acid (RNA) in primary DENV infection.

ELIGIBILITY:
Inclusion Criteria:

* Participant with a referral note/documentation from a health care facility or practitioner indicating non-structural 1 protein (NS1) positive for dengue virus (DENV), positive NS1 rapid test at pre-screening during an ambulatory visit, or participant who tests NS1 positive at the site
* Participant reported a fever with an onset within the last 48 hours
* A woman of childbearing potential must have a negative serum pregnancy test at screening
* A woman must be: a. not of childbearing potential, b. of childbearing potential and practicing a highly effective, preferably user-independent method of contraception (failure rate of less than [<] 1% per year when used consistently and correctly) and agrees to remain on a highly effective method while receiving study intervention and until at least 90 days after last dose- the end of relevant systemic exposure
* A male participant must agree not to donate sperm for the purpose of reproduction during the study and for a minimum of 90 days after receiving the last dose of study intervention

Exclusion Criteria:

* Participant with any clinical signs and symptoms for severe dengue according to the world health organization (WHO) criteria (such as severe plasma leakage leading to dengue shock syndrome [DSS], fluid accumulation with respiratory distress, severe bleeding, sever organ involvement)
* Use of any cytochrome 3A4 (CYP3A4) inducers (example, phenytoin, rifampin), UDP glucuronosyltransferase family 1 member A9 (UGT1A9) inducers (example, rifampin), or substrates for CYP3A4 with a narrow therapeutic range (example, alfentanil, cyclosporin), or sensitive breast cancer resistance protein (BCRP) substrates (example, pravastatin and folic acid) from 14 days before first dose of study drug until 28 days after last dose of study drug. Systemic use of strong CYP3A4 inhibitors (example, clarithromycin, itraconazole) or UGT1A9 inhibitors (example, probenecid, mefenamic acid) from 7 days before first dose of study drug until 28 days after last dose of study drug
* History of malignancy within 5 years before screening (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy, which is considered cured with minimal risk of recurrence)
* Had major surgery, (example, requiring general anesthesia) within 4 weeks before screening, or will not have fully recovered from surgery, or has surgery planned during the time the participant is expected to participate in the study
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunomodulation therapy such as anti-cancer chemotherapy or radiation therapy; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2022-09-24 (Actual); Study Completion 2023-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson and Johnson is available at www.janssen.com/clinical- trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Due to small number of enrolled participants, planned data collection and analysis was not performed for the efficacy objectives and no data was reported for efficacy outcome measures and thus only safety analysis data were reported.
Groups:
- JNJ-64281802: Participants received 2 initial loading dose of JNJ-64281802 up to Day 2, followed by a maintenance dose on Days 3, 4, and 5.
- Placebo: Participants received oral dose of placebo matching to JNJ-64281802 every 8 hour (q8h) and once daily on Day 4 and Day 5.
Period: Overall Study
Arm/Group | JNJ-64281802 | Placebo
Started | 2 | 3
Completed | 2 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | JNJ-64281802 | Placebo | Total
Number analyzed (Participants) | 2 | 3 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 5
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (9.9) | 37.7 (9.5) | 41.4 (9.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 3 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  SINGAPORE | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Log10-Transformed Dengue Virus (DENV) RiboNucleic Acid (RNA) Viral Load (VL) Curve From Baseline Until Day 5 (AUCD1-D5 [log10VL]).
Description: The antiviral activity of JNJ-64281802 versus placebo in terms of reduction of DENV RNA in participants with a primary DENV infection was planned to be measured by the area under the log10-transformed DENV RNA viral load concentration-time curves from baseline (Day 1) until Day 5 (AUCD1-D5 [log10VL]).
Time Frame: Baseline (Day 1) upto Day 5
Population: Due to the small number of enrolled participants, planned data collection and analysis was not performed and thus no data was reported for this outcome measure.
Arm/Group | JNJ-64281802 | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. TEAEs were those AE events that occurred at or after the initial administration of study intervention through the last onsite visit.
Time Frame: From Day 1 up to the last onsite visit (Day 30)
Population: Safety population included all randomized participants who had taken at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | JNJ-64281802 | Placebo
Number analyzed (Participants) | 2 | 3
Participants | 2 | 3

3. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Electrocardiogram (ECG) Findings
Description: Number of participants with clinically significant abnormalities in ECGs parameters as assessed based on investigator's discretion were reported.
Time Frame: From Day 1 up to the last onsite visit (Day 30)
Population: Safety population included all randomized participants who had taken at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | JNJ-64281802 | Placebo
Number analyzed (Participants) | 2 | 3
Participants | 0 | 0

4. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Physical Examination
Description: Number of participants with clinically significant abnormalities in physical examination parameters (head/neck/thyroid, eyes/ears/nose/throat, respiratory, cardiovascular, lymph nodes, abdomen, skin, musculoskeletal, and neurological) as assessed based on investigator's discretion were reported.
Time Frame: From Day 1 up to the last onsite visit (Day 30)
Population: Safety population included all randomized participants who had taken at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | JNJ-64281802 | Placebo
Number analyzed (Participants) | 2 | 3
Participants | 0 | 1

5. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Vital Signs
Description: Number of participants with clinically significant abnormalities in vital signs (temperature, pulse/heart rate, respiratory rate, peripheral capillary oxygen saturation [spO2], input-output [I/O] ratio and blood pressure) as assessed based on investigator's discretion were reported.
Time Frame: From Day 1 up to the last onsite visit (Day 30)
Population: Safety population included all randomized participants who had taken at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | JNJ-64281802 | Placebo
Number analyzed (Participants) | 2 | 3
Participants | 1 | 0

6. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Laboratory Parameters
Description: Number of participants with clinically significant abnormalities in laboratory parameters (serum chemistry, hematology, and coagulation) were reported. Clinical significance was defined as per investigator's judgement.
Time Frame: From Day 1 up to the last onsite visit (Day 30)
Population: Safety population included all randomized participants who had taken at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | JNJ-64281802 | Placebo
Number analyzed (Participants) | 2 | 3
Participants | 2 | 3

7. Secondary Outcome: Plasma Concentrations of JNJ-64281802
Description: Plasma Concentrations of JNJ-64281802 was assessed. Due to small number of enrolled participants, no summary statistics analysis was performed. Participant wise data were reported for this outcome measure.
Time Frame: Predose: 0, 8, 16 hours on Day 1; 24, 32, 40 hours on Day 2; Day 4, Day 5; and Post dose: 4, 12 hours on Day 1; 28, 36 hours on Day 2; 48 hours on Day 3; Day 6, Day 14, Day 21, Day 28
Population: Pharmacokinetic population which included all participants who receive at least 1 dose of study drug and who had at least 1 plasma concentration data value after dosing. Data for this outcome measure was not planned to be collected and analyzed for the placebo arm.
Measure: Number; unit: nanograms per milliliter
Arm/Group | JNJ-64281802
Number analyzed (Participants) | 2
nanograms per milliliter
  Participant 1: Day 1, pre-dose: number analyzed (Participants) | 1
  Participant 1: Day 1, pre-dose | 5.00
  Participant 1: Day 1, 4 hr post-dose: number analyzed (Participants) | 1
  Participant 1: Day 1, 4 hr post-dose | 1840
  Participant 1: Day 1, 8 hr pre-dose: number analyzed (Participants) | 1
  Participant 1: Day 1, 8 hr pre-dose | 2380
  Participant 1: Day 1, 12 hr post-dose: number analyzed (Participants) | 1
  Participant 1: Day 1, 12 hr post-dose | 3210
  Participant 1: Day 1, 16 hr pre-dose: number analyzed (Participants) | 1
  Participant 1: Day 1, 16 hr pre-dose | 3530
  Participant 1: Day 2, 24 hr pre-dose: number analyzed (Participants) | 1
  Participant 1: Day 2, 24 hr pre-dose | 3300
  Participant 1: Day 2, 28 hr post-dose: number analyzed (Participants) | 1
  Participant 1: Day 2, 28 hr post-dose | 3260
  Participant 1: Day 2, 32 hr pre-dose: number analyzed (Participants) | 1
  Participant 1: Day 2, 32 hr pre-dose | 3840
  Participant 1: Day 2, 36 hr post-dose: number analyzed (Participants) | 1
  Participant 1: Day 2, 36 hr post-dose | 4240
  Participant 1: Day 2, 40 hr pre-dose: number analyzed (Participants) | 1
  Participant 1: Day 2, 40 hr pre-dose | 4580
  Participant 1: Day 3, 48 hr post-dose: number analyzed (Participants) | 1
  Participant 1: Day 3, 48 hr post-dose | 4880
  Participant 1: Day 4, pre-dose: number analyzed (Participants) | 1
  Participant 1: Day 4, pre-dose | 3790
  Participant 1: Day 5, pre-dose: number analyzed (Participants) | 1
  Participant 1: Day 5, pre-dose | 3880
  Participant 1: Day 6, post-dose: number analyzed (Participants) | 1
  Participant 1: Day 6, post-dose | 4270
  Participant 1: Day 14 post-dose: number analyzed (Participants) | 1
  Participant 1: Day 14 post-dose | 1950
  Participant 1: Day 21 post dose: number analyzed (Participants) | 1
  Participant 1: Day 21 post dose | 1520
  Participant 1: Day 28 post dose: number analyzed (Participants) | 1
  Participant 1: Day 28 post dose | 954
  Participant 2: Day 1, pre-dose: number analyzed (Participants) | 1
  Participant 2: Day 1, pre-dose | 5.00
  Participant 2: Day 1, 4 hr post-dose: number analyzed (Participants) | 1
  Participant 2: Day 1, 4 hr post-dose | 694
  Participant 2: Day 1, 8 hr pre-dose: number analyzed (Participants) | 1
  Participant 2: Day 1, 8 hr pre-dose | 819
  Participant 2: Day 1, 12 hr post-dose: number analyzed (Participants) | 1
  Participant 2: Day 1, 12 hr post-dose | 1390
  Participant 2: Day 1, 16 hr pre-dose: number analyzed (Participants) | 1
  Participant 2: Day 1, 16 hr pre-dose | 1460
  Participant 2: Day 2, 24 hr pre-dose: number analyzed (Participants) | 1
  Participant 2: Day 2, 24 hr pre-dose | 1720
  Participant 2: Day 2, 28 hr post-dose: number analyzed (Participants) | 1
  Participant 2: Day 2, 28 hr post-dose | 2430
  Participant 2: Day 2, 32 hr pre-dose: number analyzed (Participants) | 1
  Participant 2: Day 2, 32 hr pre-dose | 2400
  Participant 2: Day 2, 36 hr post-dose: number analyzed (Participants) | 1
  Participant 2: Day 2, 36 hr post-dose | 3710
  Participant 2: Day 2, 40 hr pre-dose: number analyzed (Participants) | 1
  Participant 2: Day 2, 40 hr pre-dose | 3960
  Participant 2: Day 3, 48 hr post-dose: number analyzed (Participants) | 1
  Participant 2: Day 3, 48 hr post-dose | 3190
  Participant 2: Day 4, pre-dose: number analyzed (Participants) | 1
  Participant 2: Day 4, pre-dose | 1780
  Participant 2: Day 5, pre-dose: number analyzed (Participants) | 1
  Participant 2: Day 5, pre-dose | 2130
  Participant 2: Day 6, post-dose: number analyzed (Participants) | 1
  Participant 2: Day 6, post-dose | 2440
  Participant 2: Day 14 post-dose: number analyzed (Participants) | 1
  Participant 2: Day 14 post-dose | 1370
  Participant 2: Day 21 post dose: number analyzed (Participants) | 1
  Participant 2: Day 21 post dose | 991
  Participant 2: Day 28 post dose: number analyzed (Participants) | 1
  Participant 2: Day 28 post dose | 686

8. Secondary Outcome: Number of Participants With Occurrence of Detectable Dengue Virus (DENV) RiboNucleic Acid (RNA) in Primary DENV Infection
Description: Number of participants with occurrence of detectable DENV RNA in primary DENV infection was a planned analysis.
Time Frame: Predose: 24 hour on Day 2; Post dose: 12 hour on Day 1; 36 hour on Day 2; Days 3, 4, 5, 6, 7, 8, 9, 14, 21 and 28
Population: Due to small number of enrolled participants, planned data collection and analysis was not performed and thus no data was reported for this outcome measure.
Arm/Group | JNJ-64281802 | Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Time to Undetectable Dengue Virus (DENV) RiboNucleic Acid (RNA) in Primary DENV Infection
Description: Time to undetectable DENV RNA in primary DENV infection was a planned analysis.
Time Frame: Predose: 24 hour on Day 2; Post dose: 12 hour on Day 1; 36 hour on Day 2; Days 3, 4, 5, 6, 7, 8, 9, 14, 21 and 28
Population: as for outcome 8
Arm/Group | JNJ-64281802 | Placebo
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Area Under the Plasma Concentration Time Curve During One Dosing Interval (AUC[Tau]) of JNJ-64281802
Description: AUC[tau] is defined as area under the plasma concentration time curve during one dosing interval of JNJ-64281802.
Time Frame: 0, 8, 16 hours pre-dose on Day 1; 4 and 12 hours post-dose on Day 1
Population: Due to small number of enrolled participants, formal analysis was not performed for the planned PK parameters and thus no data was reported for this outcome measure
Arm/Group | JNJ-64281802
Number analyzed (Participants) | 0

11. Secondary Outcome: Trough (Pre-dose) Analyte Concentration (Ctrough) of JNJ-64281802
Description: Ctrough is defined as plasma concentration just prior to the beginning or at the end of a dosing interval of JNJ-64281802.
Time Frame: Pre-dose on Day 1: 0 hour, 8 hour, 16 hour; pre-dose on Day 2: 24 hour, 32 hour, 40 hour; pre-dose on Day 4 and Day 5
Population: as for outcome 10
Arm/Group | JNJ-64281802
Number analyzed (Participants) | 0

12. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of JNJ-64281802
Description: Cmax is defined as the maximum observed plasma concentration of JNJ-64281802.
Time Frame: 0, 8, 16 hours pre-dose on Day 1; 4 and 12 hours post-dose on Day 1
Population: as for outcome 10
Arm/Group | JNJ-64281802
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From Day 1 up to the last onsite visit (Day 30)
Description: Safety population which included all randomized participants who had taken at least 1 dose of study intervention.
Arm/Group | JNJ-64281802 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/3
Other Adverse Events (participants affected / at risk) | 2/2 | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | JNJ-64281802 (N=2) | Placebo (N=3)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2
Abdominal Distension (Gastrointestinal disorders) | 0 | 2
Abdominal Pain (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Epigastric Discomfort (Gastrointestinal disorders) | 0 | 1
Gingival Bleeding (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 3
Vomiting (Gastrointestinal disorders) | 0 | 2
Fatigue (General disorders) | 0 | 1
Covid-19 (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Viral Infection (Infections and infestations) | 0 | 1
Scratch (Injury, poisoning and procedural complications) | 0 | 1
Aspartate Aminotransferase Increased (Investigations) | 0 | 2
Lymphocyte Count Decreased (Investigations) | 1 | 0
Neutrophil Count Decreased (Investigations) | 1 | 0
Platelet Count Decreased (Investigations) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Dizziness Postural (Nervous system disorders) | 1 | 0
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1 | 2
Flushing (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Since feasibility of enrollment was impacted by COVID, sponsor terminated the study. Due to small number of enrolled participants, planned data collection and analysis was not performed for the efficacy objectives and thus no data was reported for efficacy outcome measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2022-06-06): https://cdn.clinicaltrials.gov/large-docs/80/NCT04906980/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-04): https://cdn.clinicaltrials.gov/large-docs/80/NCT04906980/SAP_001.pdf